CLINICAL TRIAL: NCT00439309
Title: Randomized Study to Evaluate Safety & Effectiveness of Vascular Sealant to Control Suture Line Bleeding
Brief Title: Study to Evaluate Safety & Effectiveness of Vascular Sealant System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAS-06-001
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VascuSeal (Experimental): Consists of two liquids that when mixed together in situ rapidly cross-link to form a biocompatible absorbable sealant that is tissue adherent. These liquids are sprayed onto tissues using the Dual Liquid Applicator. The formed Sealant remains intact for approximately 2 to 7 days. During this period the Sealant undergoes hydrolysis where it is absorbed into the circulatory system and is excreted through the kidneys.
  Interventions: Device: VascuSeal
- GELFOAM/THROMBIN (Active Comparator): GELFOAM/THROMBIN description - GELFOAM Sterile Compressed Sponge is a medical device intended for application to bleeding surfaces as a hemostatic. It is water-insoluble, off-white, nonelastic, porous, pliable product prepared from purified porcine Skin Gelatin USP Granulates and Water for Injection, USP. It may be cut without fraying and is able to absorb and hold within its interstices, many times its weight of blood and other fluids. Although not necessary, GELFOAM can be used either with or without thrombin to obtain hemostasis.
  Interventions: Device: Gelfoam/Thrombin

INTERVENTIONS:
Device: Gelfoam/Thrombin — Gelfoam/Thrombin
  Other Names: absorbable gelatin compressed sponge
  Arms: GELFOAM/THROMBIN
Device: VascuSeal — VascuSeal
  Other Names: Vascular Sealant System
  Arms: VascuSeal

SUMMARY:
To evaluate a new vascular sealant compared to control for the control of suture line bleeding after vascular reconstructive surgery.

DETAILED DESCRIPTION:
Vascular surgery encompasses a wide range of surgical procedures. In these procedures reduction of blood loss and creation of suture line is of utmost importance to the surgeon. Bleeding at the suture line may require transfusion, as well as prolonged operative and anesthesia time. Suture hole bleeding is common following using synthetic and biological grafts for vascular repair. Several topical hemostatic ans sealing agents have been developed to control suture line bleeding. This new vascular sealant possess high bonding properties, minimal tissue reaction, is biodegradable and absorbed by the body quickly. The primary focus of this study is to compare the safety and effectiveness of the vascular sealant with standard of care methods used today, specifically gelfoam/thrombin and sponge like material.

ELIGIBILITY:
Inclusion Criteria:

Subject was > 18 years of age. Scheduled for elective vascular surgery that entails placement of a PTFE vascular graft including extra-anatomic, infrainguinal bypass, and primary and secondary arteriovenous access procedures. Subject was willing and able to comply with all aspects of the treatment and evaluation schedule. Informed of the nature of the study, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site

Exclusion Criteria:

Subject had a known local or systemic infection. Subjects with known coagulopathies including hemophilia, factor deficiencies, platelet count < 80,000 u/mL, heparin induced thrombocytopenia or uncorrected INR > 1.5. Subject was participating in a clinical trial that requires treatment with another investigational device or drug. Subject was lactating or pregnant, or does not agree to use contraception for the duration of the study. Subject had a known hypersensitivity to any components of bovine thrombin preparations and/or material of bovine origin. The investigator determined that the subject should not be included in the study for reason(s) not already specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Scerbin, Study Director — Confluent Surgical
Locations (1):
- Confluent Surgical, Inc., Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled between 6APR07 & 20MAY08 at: U. Hospitals of Cleveland; Cleveland Clinic; Medical U. of Ohio Toledo; Boston Medical Center; OHSU; Southern Illinois U.; Washington Hospital Center; Penn State Heart & Vascular Inst., Georgetown U.; Brigham & Women's; Methodist Hospital; Vascular & Transplant Specialists; St. Vincent's East
Period: Treatment
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Started | 54 | 15
Completed | 54 | 15
Not Completed | 0 | 0
Period: Follow-Up
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Started | 54 | 15
Completed | 51 | 13
Not Completed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Late response by subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VascuSeal | GELFOAM/THROMBIN | Total
Number analyzed (Participants) | 54 | 15 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 11 | 41
  >=65 years | 24 | 4 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.45 (11.773) | 60.91 (12.958) | 62.51 (11.904)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 8 | 35
  Male | 27 | 7 | 34
Region of Enrollment [Number; unit: participants]
  United States | 54 | 15 | 69

OUTCOME MEASURES:

1. Primary Outcome: Sealing Success
Description: The primary effectiveness endpoint is sealing success defined as complete anastomotic suture line sealing within 10 minutes following restoration of blood flow without use of an adjunctive hemostatic technique different from the assigned treatment. The primary effectiveness endpoint was evaluated on a per subject basis. For subjects with two treated sites, the subject is considered a success only if there is complete anastomotic suture line sealing within 10 minutes at both sites.
Time Frame: Within 10 minutes following restoration of blood flow
Population: The primary effectiveness endpoint was evaluated on a per subject basis. For subjects with two treated sites, the subject is considered a success only if there is complete anastomotic suture line sealing within 10 minutes at both sites.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Number analyzed (Participants) | 54 | 15
percentage of participants | 90.7 [79.7 to 96.9] | 86.7 [59.5 to 98.3]
Statistical Analysis 1: Comparison: VascuSeal vs GELFOAM/THROMBIN; The effectiveness analyses were performed on the ITT population; Test type: Non-Inferiority or Equivalence — The sealing success rates for the investigational group and control groups were assumed to be 0.85 (85%) and 0.75 (75%), respectively, and the non-inferiority margin (10%) is 0.10. For safety reasons it was desired to have at least 100 Vascular Sealant treated subjects. It was determined that a sample size of at least 31 evaluable subjects is required for the control group. For blocking purposes, the number of evaluable control group subjects was set to 33, for a 3:1 randomization; p = 0.072, Z-Test; one-sided Z-test based on the normal approximation to the binomial distribution testing

2. Secondary Outcome: Proportion of Immediate Sealing Success at Treated Anastomoses (Anastomoses Level)
Description: A site with no suture line bleeding after blood flow is restored and monitored for a minimum period of 60 seconds to confirm cessation of blood flow
Time Frame: 60 seconds post restoration of blood flow
Measure: Number; unit: percentage of anastomotic sites
Units Other Than Participants: Anastomosis
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Number analyzed (Participants) | 54 | 15
Number analyzed (Anastomosis) | 68 | 19
percentage of anastomotic sites | 51.5 | 10.5
Statistical Analysis 1: Comparison: VascuSeal vs GELFOAM/THROMBIN; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; p-value for superiority of the Vascular Sealant System compared to the GELFOAM Treatment from two-sided test based on the GEE regression model

3. Secondary Outcome: Proportion of Overall Sealing Successes at Treated Anastomoses (Anastomoses Level)
Description: as for outcome 2
Time Frame: Within 10 minutes post restoration of blood flow
Measure: Number; unit: percentage of anastomitic sites
Units Other Than Participants: Anastomosis
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Number analyzed (Participants) | 54 | 15
Number analyzed (Anastomosis) | 68 | 19
percentage of anastomitic sites | 92.6 | 89.5
Statistical Analysis 1: Comparison: VascuSeal vs GELFOAM/THROMBIN; Test type: Superiority or Other; p = 0.654, t-test, 2 sided; p-value for superiority of the Vascular Sealant System compared to the GELFOAMTreatment from two-sided test based on the GEE regression model

4. Secondary Outcome: Time to Hemostasis
Description: Time to hemostasis determined from time circulation restored after treatment application until bleeding stopped (assessed at intervals of immediate, 1, 3, 5, 7.5 and 10 min). For subject with two sites, time to hemostasis of both sites used for analysis. Subjects for whom bleeding had not stopped within 10 min considered censored observations.
Time Frame: Within 10 minutes post restoration of blood flow
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Number analyzed (Participants) | 54 | 15
Minutes | 1.0 [0.0 to 3.0] | 5.0 [3.0 to 7.5]
Statistical Analysis 1: Comparison: VascuSeal vs GELFOAM/THROMBIN; Test type: Superiority or Other; p = 0.089, t-test, 2 sided

5. Secondary Outcome: Time to Wound Closure
Description: Time to wound closure was defined as the elapsed time between initial clamp removal at the last anastomotic site until skin closure. This endpoint was analyzed using the log-rank test to compare the two treatment groups. The Kaplan-Meier method was used to obtain estimated median times to wound closure and the corresponding 95% confidence intervals for each treatment group.
Time Frame: From initial clamp removal at the last anastomotic site until skin closure
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Number analyzed (Participants) | 54 | 15
Minutes | 53.5 [43.0 to 59.0] | 42.5 [37 to 75.0]
Statistical Analysis 1: Comparison: VascuSeal vs GELFOAM/THROMBIN; Test type: Superiority or Other; p = 0.404, Log Rank; Kaplan-Meier method was used to obtain estimated median times to wound closure and the corresponding 95% confidence intervals for each treatment group

ADVERSE EVENTS:
Time Frame: 30 days post randomization
Description: For other adverse events, adverse events were only collected with regard to the affected organ system.
Arm/Group | VascuSeal | GELFOAM/THROMBIN
Serious Adverse Events (participants affected / at risk) | 19/54 | 3/15
Other Adverse Events (participants affected / at risk) | 37/54 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VascuSeal (N=54) | GELFOAM/THROMBIN (N=15)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Arteriovenous Graft Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Incision Site Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Incision Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 2 (2) | 0 (0)
Arteriovenous Graft Thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Graft Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laboratory test Abnormal (Investigations) | 1 (1) | 0 (0)
Essential Thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial Thrombosis Limb (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VascuSeal (N=54) | GELFOAM/THROMBIN (N=15)
Blood and Lymphatic System Disorder (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Cardiac Disorder (Cardiac disorders) | 1 (1) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 5 (5) | 1 (1)
General Disorder and Administration Site Conditions (General disorders) | 8 (8) | 2 (2)
Infection and Infestation (Infections and infestations) | 4 (4) | 0 (0)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
Investigations (Investigations) | 3 (3) | 3 (3)
Metabolism and Nutrition (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Respiratroy, Thoracic And mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Vascular Disorders (Vascular disorders) | 5 (5) | 1 (1)
Nervous System Disorders (Nervous system disorders) | 1 (1) | 1 (1)
Surgical and medical Procedures (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less